CLINICAL TRIAL: NCT01413282
Title: Better Evaluation of Acute Chest Pain With Computed Tomography Angiography - A Randomized Controlled Trial
Brief Title: Better Evaluation of Acute Chest Pain With Computed Tomography Angiography
Acronym: BEACON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Koen Nieman, Associate professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BEACON-11
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Acute Coronary Syndrome; Acute Chest Pain
Keywords: Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiac CT (Active Comparator): Triage based on cardiac CT results.
  Interventions: Radiation: Cardiac CT
- Standard Care (No Intervention): Standard diagnostic management according to the European guidelines.

INTERVENTIONS:
Radiation: Cardiac CT — Calcium scan and CT coronary angiography
  Arms: Cardiac CT

SUMMARY:
The purpose of this study is to determine whether cardiac CT can improve triage of acute chest pain patients in the emergency department.

DETAILED DESCRIPTION:
Myocardial infarction remains one of the most important causes of death and disability. Therefore it is important that individuals with acute chest pain are accurately assessed without delaying appropriate treatment. Acute coronary syndrome is only one cause for sudden chest pain, which is a very common complaint in the ER. Other life threatening causes such as pulmonary embolism and aortic dissection may also be the cause, although most chest discomfort has a benign reason (musculoskeletal, hyperventilation, oesophageal reflux, etc).

The current work-up of suspected acute coronary syndrome, based on presentation, symptoms, ECG and biomarkers, is not efficient and results in unnecessary diagnostics and hospital admissions, as well as errors or delayed diagnoses, in a substantial number of patients. Computed tomography angiography (CTA) images atherosclerosis, coronary obstruction as well as myocardial hypoperfusion. We hypothesize that early use of CTA is of incremental value and allows for accurate and immediate triage of patients with acute chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Acute chest pain or equivalent
* Patients older than 30 years
* Males < 75 years and Females < 80 years

Exclusion Criteria:

* STEMI
* Troponin > 0.1
* History of known myocardial infarction, PCI or CABG
* Pregnancy
* Contrast allergy
* Renal disfunction
* No informed consent possible
* No follow-up possible

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Successful discharge rate | 30 days
  The proportion of patients discharged home without major adverse events during the following 30 days. Major adverse events are cardiovascular death or non-fatal myocardial infarction.
Diagnostic yield of invasive angiography | 30 days
  Number of patients identified with severe coronary artery disease identified by invasive angiography requiring revascularisation according to the international guidelines.

SECONDARY OUTCOMES:
Successful discharge rate for all adverse events | 30 days
  The proportion of patients discharged home without any adverse events during the following 30 days. Adverse events are cardiovascular death, non-fatal myocardial infarction, unstable angina, coronary revascularization, repeat hospital visits for chest pain.
Major adverse events | 6 months
  Composite endpoint of major adverse cardiac events at 6 months: cardiovascular death, non-fatal myocardial infarction, unstable angina, coronary revascularisation and repeat hospital visits for chest pain.
Acute coronary syndrome | Index hospital visit
  Diagnosis of acute coronary syndrome, according to international guidelines, at time of discharge.
Missed myocardial infarctions | 2 days
  Missed myocardial infarctions, at 2-day follow-up, in patients discharged from the emergency department.
Duration of hospital stay | Index hospital visit
  Duration of hospital stay
Direct medical cost | 30 days
  Direct medical costs until 30th day after ED visit.
Radiation exposure | 6 months
  Cumulative medical radiation exposure at 6 months.
Renal function | 2 days
  Change in renal function after 2 days.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Nieman, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dedic A, Lubbers MM, Schaap J, Lammers J, Lamfers EJ, Rensing BJ, Braam RL, Nathoe HM, Post JC, Nielen T, Beelen D, le Cocq d'Armandville MC, Rood PP, Schultz CJ, Moelker A, Ouhlous M, Boersma E, Nieman K. Coronary CT Angiography for Suspected ACS in the Era of High-Sensitivity Troponins: Randomized Multicenter Study. J Am Coll Cardiol. 2016 Jan 5;67(1):16-26. doi: 10.1016/j.jacc.2015.10.045. PMID 26764061